CLINICAL TRIAL: NCT06995833
Title: Durvalumab With or Without Olaparib in Patients With Endometrial Cancers Regulatory Post Marketing Surveillance
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9102R00001
Record Dates: First submitted 2025-05-28; First posted 2025-05-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives of this study are to assess the safety and effectiveness of Durvalumab with or without Olaparib (hereinafter "the study drug") in a real world setting in patients who are prescribed with the study drug under the approved indication in Korea.

This is a multicenter, prospective, observational, real world treatment study. Patients treated as part of routine practice at Korean healthcare centers by investigators will be identified and considered for inclusion in the study. The period of this study is expected to run for 4 years from the approval date of the indication for this study. Approximately 50 patients are expected to be enrolled during the study.

Patient will be followed for approximately 12 months from the first dose or up to 90 days after treatment discontinuation if the study drug is administered for less than 12 months, unless they withdraw consent, are lost to follow-up or death.

DETAILED DESCRIPTION:
Primary Objective: To assess the safety of the study drug in patients prescribed with the study drug under the approved indication(s) in Korea

Secondary Objective: To assess effectiveness of the study drug in patients prescribed with the study drug under the approved indication(s) in Korea

Exploratory Objective: To assess the safety and effectiveness of the study drug in patients prescribed with the study drug under the approved indication(s) in Korea by treatment/ MMR status

ELIGIBILITY:
Inclusion Criteria:

1. Patients eligible for the study drug according to the approved label in Korea
2. Provision of a signed and dated written informed consent by the patient or their legally acceptable representative

Exclusion Criteria:

1. Participation in any concurrent interventional trials during the period of the study drug treatment
2. Other off-label indications according to the approved label in Korea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be enrolled by a total surveillance method. In principle, patients treated with study drugs in accordance with local prescribing information are eligible for enrollment in this study. Each patient must meet all of the inclusion criteria and none of the exclusion criteria. Investigators should enroll the patients who initiate or are receiving treatment with study drugs after the contract date.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events (AEs), serious AEs (SAEs), adverse drug reactions (ADRs), serious ADRs (SADRs), unexpected AEs/ADRs) | Patient will be followed for approximately 12 months from the first dose or up to 90 days after treatment discontinuation if the study drug is administered for less than 12 months, unless they withdraw consent, are lost to follow-up or death.
  To assess safety of the study drugs for patients treated with the study drugs under the approved indication in Korea

SECONDARY OUTCOMES:
Real-world Progression free survival (rwPFS) | Data obtained up until progression, or the last evaluable assessment (up to 12 month +/- 30 days) in the absence of progression, will be included in the assessment of rwPFS.
  To assess effectiveness of the study drugs for patients treated with the study drugs under the approved indication in Korea

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/